CLINICAL TRIAL: NCT03845348
Title: Đánh giá hiệu quả điều trị viêm da dầu ở đầu của dầu gội Thái Dương 3 và Thái Dương 7 (A Randomized, Double Blind, Placebo Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy Shampoos TD03 and TD07 in Scalp Diseases)
Brief Title: To Evaluate the Efficacy and Safety of Shampoo TD03 and TD07 in Scalp Diseases
Acronym: TD0307
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sao Thai Duong Joint Stock Company (Industry)
Collaborators: Big Leap Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TD0307.03
Record Dates: First submitted 2019-01-10; First posted 2019-02-19 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-06

CONDITIONS: Scalp Dermatitis
MeSH Terms: interventions — Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TD3 (Experimental): TD3, bi-daily x 4 weeks
  Interventions: Other: TD03
- TD7 (Experimental): TD7, bi-daily x 4 weeks
  Interventions: Other: TD07
- Ketoconazole 2% (Active Comparator): Ketoconazole 2% shampoo bi-daily x 4 weeks
  Interventions: Drug: Ketoconazole 2% Shampoo

INTERVENTIONS:
Other: TD03 — Shampoo TD 3 days
  Arms: TD3
Other: TD07 — Shampoo TD 7 days
  Arms: TD7
Drug: Ketoconazole 2% Shampoo — Ketoconazole 2% Shampoo
  Arms: Ketoconazole 2%

SUMMARY:
Scalp Conditions are common chronic skin inflamations with the occurence rate of 1 - 5 % among the population. TD03 shampoo and TD07 shampoo are widely used to avoid hair loss with successful rate reaching nearly 95%. This trial is going to evaluate the efficacy of getting rid of dandruff as well as the safety of the investigational products in comparison to a reference (ketoconazole 2%) during a 4-week treatment period.

DETAILED DESCRIPTION:
Scalp Conditions are common chronic skin inflamations with the occurence rate of 1 - 5 % among the population. TD03 shampoo and TD07 shampoo are widely used to avoid hair loss with successful rate reaching nearly 95%. With herbal ingredients including Gleditsia, Morus alba, Ocimum tenuiflorum, Oroxylum indicum, Ageratum conyzoides, the investigational products could reduce the severity of inflamation, infection and help to prevent hair loss. This trial is planning to evaluate the efficacy of the IPs in terms of inflamation reduction, dandruff reduction on subjects using the IPs compared to a reference (ketoconazole 2%).

The trial is intended to last for 18 months with subject visits and 3 arms (122 subjects per arm). The first arm receive TD3 while TD7 is provided to the second arm in comparison to the placebo of the last arm. It will be conducted at National Hospital of Dermato - Venerology, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old and signed the ICF.
* Diagnosed with head skin inflamtion with IGA <= 3.
* Voluntary sign the ICF before any procedures.
* No hypersentivity to the IP.

Exclusion Criteria:

* Use oral antifungal 1 month prior to the trial participation or topical antifungal 2 weeks prior to the trial participation.
* Suffering chronic or acute diseases that may affect the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in IGA scale at 4 week-treatment | 4 weeks
  Change from baseline in IGA scale at 4 week-treatment of TD3 and TD7 compared to that of Ketoconazole 2% shampoo.
The numbers of subjects with AE/SAE | 4 weeks
  The numbers of subjects with AE/SAE as defined in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Phuong TM Pham, Principal Investigator — National Hospital of Dermatology
Locations (1):
- Nationa Hospital of Dermatology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No